CLINICAL TRIAL: NCT05752435
Title: Comparison of Therapeutic Efficacy Between Intralesional Bleomycin and Cryotherapy in Plantar Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Siddiqui, Head of Department of Dermatology, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMHAbbottabad-Derma
Record Dates: First submitted 2023-02-01; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Viral Wart
MeSH Terms: conditions — Warts | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial (RCT)
Who Masked: Outcomes Assessor
Masking Description: cure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLEOMYCIN (Active Comparator): COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS
  Interventions: Procedure: COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS
- CRYOTHERAPY (Active Comparator): COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS
  Interventions: Procedure: COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS

INTERVENTIONS:
Procedure: COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS — comparison of therapeutic efficacy between intralesional bleomycin and cryotherapy in plantar warts

SUMMARY:
A randomized control trial to compare the efficacy difference between intralesional bleomycin and cryotherapy in treating plantar warts.

DETAILED DESCRIPTION:
In spite of many available studies on bleomycin and cryotherapy in treating warts, little head-to-head research is carried out to compare the efficacy of these treatments. This study shows clear difference in the clearance of warts treated with intralesional bleomycin and cryotherapy.

ELIGIBILITY:
Inclusion Criteria

-healthy individuals of both genders between 18 to 50 years

Exclusion Criteria

* Pregnant and Lactating women
* history of vascular diseases/ chilblains
* Immunocompromised patients
* Treated previously for warts

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
comparative effecacy of intra lesional bleomycin vs cryotherapy in treating plantar warts within 30 days of treatment | 30 days of treatment
  Intralesional bleomycin is more effective than cryotherapy in treating plantar warts within

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Dr Siddiqui, FCPS, Study Director — Combined Military Hospital Abbottabad
Locations (1):
- Adeel Siddiqui, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: COMPARISON OF THERAPEUTIC EFFICACY BETWEEN INTRALESIONAL BLEOMYCIN AND CRYOTHERAPY IN PLANTAR WARTS
Access Criteria: via email